CLINICAL TRIAL: NCT07225114
Title: Academic-Industrial Partnership for Translation of Acoustic Angiography: Contrast Enhanced Super Resolution (CESR) Imaging
Brief Title: Translation of Acoustic Angiography: Contrast Enhanced Super Resolution (CESR) Imaging
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: LCCC2451; R01CA220681 (NIH)
Record Dates: First submitted 2025-11-03; First posted 2025-11-05 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer; Kidney Neoplasms; Liver Neoplasms
Keywords: Definity®; perflutren lipid; healthy volunteers; ultrasound; cross-sectional imaging
MeSH Terms: conditions — Breast Neoplasms; Kidney Neoplasms; Liver Neoplasms | interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Arm 1: Healthy Volunteers (Experimental): Participants without any disease diagnosis.
  Interventions: Drug: contrast agent perflutren lipid; Device: Ultrasound Imaging
- Arm 2: Breast Imaging Patients (Experimental): Participants are going to be assessed breast cancer.
  Interventions: Drug: contrast agent perflutren lipid; Device: Ultrasound Imaging
- Arm 3: Kidney Imaging Patients (Experimental): Participants are going to be assessed kidney cancer.
  Interventions: Drug: contrast agent perflutren lipid; Device: Ultrasound Imaging
- Arm 4: Liver Imaging Patients (Experimental): Participants are going to be assessed liver cancer.
  Interventions: Drug: contrast agent perflutren lipid; Device: Ultrasound Imaging

INTERVENTIONS:
Drug: contrast agent perflutren lipid — At the time of imaging, the contrast agent perflutren lipid will be administered, intravenous (IV). All patients will be visually monitored for signs or symptoms of a contrast administration reaction once the drug is administered for a 15-minute period.
Device: Ultrasound Imaging — Contrast Enhanced Super Resolution (CESR) imaging involves a research ultrasound scanner as well as conventional b-mode ultrasound to guide the location of the imaging. The conventional ultrasound will be conducted just prior to CESR imaging for localization.
  Other Names: Contrast Enhanced Super Resolution (CESR)

SUMMARY:
This is a 4-arm, single-center study involving 40 participants. Ten healthy volunteers will be enrolled for system imaging optimization, and thirty (30) patients with previously identified lesions in the breast, liver, or kidney-based on prior ultrasound or cross-sectional imaging-will be imaged. Recruitment will be conducted such that ten patients are included from each anatomic region.

The fourth arm will consist of 10 healthy volunteers who will be imaged to allow optimization of imaging parameters. Optimization is is required again due to the use of a different ultrasound system employing a new imaging technique. Parameters such as frame rate, power, depth of imaging, and linear translation rate will be adjusted during this process.

The primary objectives of the study are to assess the sensitivity and specificity of Contrast Enhanced Super-Resolution (CESR) imaging in evaluating known lesions in the breast, liver, and kidney. These results will be compared with pathological findings. The secondary objectives are to compare the sensitivity and specificity of CESR imaging with those of traditional B-mode ultrasound in differentiating malignant from benign lesions in these same organs.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years old
* Patient had a diagnostic ultrasound study performed at University of North Carolina
* Scheduled for a biopsy
* Lesion visualized on ultrasound
* Able to provide informed consent
* Negative urine pregnancy test in women of child-bearing potential

Exclusion Criteria:

* Institutionalized subject (prisoner or nursing home patient)
* Critically ill or medically unstable and whose critical course during the observation period would be unpredictable (e.g., chronic obstructive pulmonary disease (COPD)
* Known hypersensitivity to sulfur hexafluoride or to any component of perflutren lipid (Definity®)
* Active cardiac disease including any of the following
* Severe congestive heart failure (class IV in accordance with the classification of the New York Heart Association)
* Unstable angina.
* Severe arrhythmia (i.e., ventricular tachycardia, flutter fibrillation; ventricular premature complexes occurring close to the preceding T-wave, multifocal complexes).
* Myocardial infarction within 14 days prior to the date of proposed Definity® administration.
* Pulmonary hypertension
* Cardiac shunts

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 40 (Estimated)
Dates: Start 2025-11-04 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of Contrast Enhanced Super-Resolution (CESR) breast imaging | Biopsy date (Up to 2 months)
  Sensitivity of Contrast Enhanced Super-Resolution (CESR) breast imaging will be evaluated by comparing image analyses to the pathological results for these lesions.
  Sensitivity will be defined as the proportion of lesions detected by CESR to be positive among lesions confirmed as positive by pathological results.
Specificity of Contrast Enhanced Super-Resolution (CESR) breast imaging | Biopsy date (Up to 2 months)
  Specificity of Contrast Enhanced Super-Resolution (CESR) breast imaging will be evaluated by comparing image analyses to the pathological results for these lesions.
  Specificity will be defined as the proportion of lesions detected by CESR to be negative among lesions confirmed as negative by pathological results.
Sensitivity of Contrast Enhanced Super-Resolution (CESR) kidney imaging | Biopsy date (Up to 2 months)
  Sensitivity of Contrast Enhanced Super-Resolution (CESR) kidney imaging will be evaluated by comparing image analyses to the pathological results for these lesions.
  Sensitivity will be defined as the proportion of lesions detected by CESR to be positive among lesions confirmed as positive by pathological results.
Specificity of Contrast Enhanced Super-Resolution (CESR) kidney imaging | Biopsy date (Up to 2 months)
  Specificity of Contrast Enhanced Super-Resolution (CESR) kidney imaging will be evaluated by comparing image analyses to the pathological results for these lesions.
  Specificity will be defined as the proportion of lesions detected by CESR to be negative among lesions confirmed as negative by pathological results.
Sensitivity of Contrast Enhanced Super-Resolution (CESR) liver imaging | Biopsy date (Up to 2 months)
  Sensitivity of Contrast Enhanced Super-Resolution (CESR) liver imaging will be evaluated by comparing image analyses to the pathological results for these lesions.
  Sensitivity will be defined as the proportion of lesions detected by CESR to be positive among lesions confirmed as positive by pathological results.
Specificity of Contrast Enhanced Super-Resolution (CESR) liver imaging | Biopsy date (Up to 2 months)
  Specificity of Contrast Enhanced Super-Resolution (CESR) liver imaging will be evaluated by comparing image analyses to the pathological results for these lesions.
  Specificity will be defined as the proportion of lesions detected by CESR to be negative among lesions confirmed as negative by pathological results.

SECONDARY OUTCOMES:
Comparison of Contrast Enhanced Super-Resolution (CESR) imaging with traditional b-mode ultrasound- breast | Biopsy date (Up to 2 months)
  The sensitivity and specificity of CESR imaging with traditional b-mode ultrasound will be compared in the distinction of malignant versus benign breast lesions.
Comparison of Contrast Enhanced Super-Resolution (CESR) imaging with traditional b-mode ultrasound- kidney | Biopsy date (Up to 2 months)
  The sensitivity and specificity of CESR imaging with traditional b-mode ultrasound will be compared in the distinction of malignant versus benign kidney lesions.
Comparison of Contrast Enhanced Super-Resolution (CESR) imaging with traditional b-mode ultrasound- liver | Biopsy date (Up to 2 months)
  The sensitivity and specificity of CESR imaging with traditional b-mode ultrasound will be compared in the distinction of malignant versus benign liver lesions.

CONTACTS AND LOCATIONS:
Overall Officials: Yueh Lee, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- The University of North Carolina, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: University of North Carolina Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials